CLINICAL TRIAL: NCT01122589
Title: Sustaining Tobacco Abstinence After Incarceration
Brief Title: Working Inside for Smoking Elimination
Acronym: WISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Memorial Hospital of Rhode Island (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Jennifer G. Clarke, MD MPH, Memorial Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WISE 09-21; 1R01DA024093-01A2 (NIH)
Record Dates: First submitted 2010-05-12; First posted 2010-05-13 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Cigarette Smoking; Tobacco Smoking
Keywords: Smoking Abstinence; Smoking Cessation
MeSH Terms: conditions — Cigarette Smoking; Tobacco Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivation Interviewing/CBT (Experimental)
  Interventions: Behavioral: Motivational Interviewing/CBT
- Control (Active Comparator): Receive a smoking cessation pamphlet and watch a series of six weekly 30-45 minutes general wellness videos.
  Interventions: Other: CONcise Tapes Reviewing Obstacles to healthy Living (CONTROL)

INTERVENTIONS:
Behavioral: Motivational Interviewing/CBT — 6 sessions of in jail MI/CBT counseling will be administered.
  Arms: Motivation Interviewing/CBT
Other: CONcise Tapes Reviewing Obstacles to healthy Living (CONTROL) — a series of six weekly 30-45 minutes general wellness videos
  Arms: Control

SUMMARY:
The purpose of this study is to determine the extent to which an Intentional Behavioral Intervention will increase tobacco quit rates post release among incarcerated men and women.

DETAILED DESCRIPTION:
Quitting smoking reduces the risks of developing smoking related illnesses as well as the morbidity and mortality associated with these illnesses. In 2006 approximately 44.5 million American adults smoked an overall prevalence of 20.8%. The prevalence is much higher among incarcerated populations and approximately 80% of the women in RI smoked prior to incarceration. This proposal is designed to evaluate an intervention utilizing Motivational Interviewing (MI) and Cognitive Behavioral Therapy (CBT) to provide the skills necessary to maintain smoking abstinence after release. MI utilizes specific techniques for providing feedback on an individual's risk and self efficacy. CBT provides the skills necessary to maintain abstinence after release. The investigators plan to recruit 350 men and women from the Rhode Island Department of Corrections and randomize them to two interventions: an Intentional Behavioral Intervention (IBI) with 6 sessions of in jail MI/CBT and two post release booster sessions compared to CONcise Tapes Reviewing Obstacles to healthy Living (CONTROL) group which will receive a smoking cessation pamphlet and watch a series of six weekly 30-45 minutes general wellness videos.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Daily smokers over the past 30 non-institutionalized days (prior to Incarceration)
* Expected place of residence after release within 15 miles of follow-up site
* Agree to participate in the study protocol and be available within one month post release
* Speak English
* Provides at least two pieces of locator information
* Scheduled to be released within eight weeks

Exclusion Criteria:

* Inability to give informed consent secondary to organic brain function, not having own legal guardianship, or active psychosis or otherwise not able to participate in the intervention or assessments (deaf, blind, or impaired communication skills that impair ability to participate in computerized assessment or counseling)
* Housed in a segregation unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-04 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Smoking abstinence | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer G Clarke, MD, Principal Investigator — Memorial Hospital of Rhode Island
Locations (1):
- Memorial Hospital of Rhode Island, Pawtucket, Rhode Island, United States

REFERENCES:
- [Derived] van den Berg JJ, Roberts MB, Bock BC, Martin RA, Stein LA, Parker DR, McGovern AR, Shuford SH, Clarke JG. Changes in Depression and Stress after Release from a Tobacco-Free Prison in the United States. Int J Environ Res Public Health. 2016 Jan 12;13(1):114. doi: 10.3390/ijerph13010114. PMID 26771622
- [Derived] Parker DR, Roberts MB, van den Berg JJ, Bock B, Stein LA, Martin RA, Clarke JG. Exploration of Incarcerated Men's and Women's Attitudes of Smoking in the Presence of Children and Pregnant Women: Is There a Disparity Between Smoking Attitudes and Smoking Behavior? Nicotine Tob Res. 2016 May;18(5):919-25. doi: 10.1093/ntr/ntv112. Epub 2015 May 25. PMID 26014453
- [Derived] Clarke JG, Martin SA, Martin RA, Stein LA, van den Berg JJ, Parker DR, McGovern AR, Roberts MB, Bock BC. Changes in smoking-related symptoms during enforced abstinence of incarceration. J Health Care Poor Underserved. 2015 Feb;26(1):106-18. doi: 10.1353/hpu.2015.0014. PMID 25702731
- [Derived] Clarke JG, Stein LA, Martin RA, Martin SA, Parker D, Lopes CE, McGovern AR, Simon R, Roberts M, Friedman P, Bock B. Forced smoking abstinence: not enough for smoking cessation. JAMA Intern Med. 2013 May 13;173(9):789-94. doi: 10.1001/jamainternmed.2013.197. PMID 23567902
- [Derived] Clarke JG, Martin RA, Stein L, Lopes CE, Mello J, Friedmann P, Bock B. Working Inside for Smoking Elimination (Project W.I.S.E.) study design and rationale to prevent return to smoking after release from a smoke free prison. BMC Public Health. 2011 Oct 5;11:767. doi: 10.1186/1471-2458-11-767. PMID 21974746